CLINICAL TRIAL: NCT04550338
Title: Antiviral Effects of Tranexamic Acid (TXA) as a Preventative Treatment Following COVID-19 Exposure
Brief Title: Antiviral Effects of TXA as a Preventative Treatment Following COVID-19 Exposure
Acronym: TXACOVIDPREV
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: With vaccination efforts ongoing, a feasibility survey indicated there would be inadequate recruitment
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Timothy Ness, MD, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TXA.COVID.3
Record Dates: First submitted 2020-09-13; First posted 2020-09-16 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: COVID-19
Keywords: COVID-19; tranexamic acid; preventative therapy; prophylactic therapy
MeSH Terms: conditions — COVID-19 | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, double-blind, randomized, controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Once patient is consented, pharmacy will randomize to one of two arms and prepare coded sets of drugs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tranexamic Acid Treatment (Experimental)
  Interventions: Drug: Tranexamic acid
- Placebo Treatment (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic acid — Oral administration of blinded medications
  Arms: Tranexamic Acid Treatment
Drug: Placebo — Oral administration of blinded medications
  Arms: Placebo Treatment

SUMMARY:
A recent report in Physiolological Reviews proposed that the endogenous protease plasmin acts on SARS-CoV-2 by cleaving a newly inserted furin site in the S protein portion of the virus resulting in increased infectivity and virulence. A logical treatment that might blunt this process would be the inhibition of the conversion of plasminogen to plasmin. Fortunately, there is an inexpensive, commonly used drug, tranexamic acid, TXA, which suppresses this conversion and could be re-purposed for the treatment of COVID-19. TXA is a synthetic analog of the amino acid lysine which reversibly binds four to five lysine receptor sites on plasminogen. This reduces conversion of plasminogen to plasmin, and is normally used to prevent fibrin degradation. TXA is FDA approved for the outpatient treatment of heavy menstrual bleeding (typical dose 1300 mg p.o. TID x 5 days) and off-label use for many other indications. TXA is used perioperatively as a standard-of-care at UAB for orthopedic and cardiac bypass surgeries. It has a long track record of safety such that it is used over-the-counter in other countries as an antiviral and for the treatment of cosmetic dermatological disorders. Given the potential benefit and limited toxicity of TXA it would appear warranted to perform randomized, double-blind placebo controlled exploratory trial at UAB as a prophylactic antiviral treatment following exposure to COVID-19 in order to determine whether it reduces infectivity and virulence of the SARS-CoV-2 virus as hypothesized. Involvement of each patient is only for 7 days before primary endpoints and 30 days for final data collection.

DETAILED DESCRIPTION:
Patients who are self-identified as having had close personal contact with an individual who has tested positive for COVID-19 will be invited to enroll in the study. On Day 1 they will be consented and randomized to one of two arms of the study: Arm 1 will consist of a 5 day treatment with tranexamic acid (TXA; 1300 mg p.o. TID x 5 days) and Arm 2 will consist of a 5 day treatment with an identical appearing placebo. All subjects will be tested using nasopharyngeal RNA swabs for the presence of the SARS-CoV-2 virus on Days 1 and 7. The primary endpoint will be conversion from a negative test for COVID-19 on Day 1, to a positive test on Day 7. Secondary data related to symptoms and co-morbidities will also be gathered.

Subjects who are positive for COVID-19 on Day 1 will not be included in the primary endpoint analysis for this study, but will receive the same 5 days of treatment and their data used for secondary analyses including safety.

All subjects in Arm 1 will also be treated with apixaban (5 mg p.o. BID x 5 days) to mitigate potential risks associated with hypercoagulability which have been noted in COVID-19 patients and which could be made worse with TXA treatment. The subjects in Arm 2 who received placebo in place of TXA will receive a second placebo tablet in place of apixaban.

Patients will be consented via the existent mechanisms associated with outpatient recruitment for all COVID-related studies at UAB. Consent would be performed remotely. All nasopharyngeal swabs will be obtained through the existent mechanisms for COVID-19 testing at UAB. Follow-up would consist of daily phone/internet contact for 7 days unless subjects acquire symptoms consistent with COVID-19, in which case they will be followed until resolution of their symptoms or for a maximum of 30 days.

ELIGIBILITY:
Inclusion Criteria:

* self-reported close exposure to individuals who test positive for COVID-19 virus

Exclusion Criteria:

* pregnancy, allergy to study drugs, history of hypercoagulability or hypocoagulability, use of anticoagulant medications, seizures, presence of intravascular stents or other instrumentation that may lead to the formation of blood clots

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Conversion from negative to positive COVID-19 test | Repeat testing after 7 days
  RNA testing of nasopharyngeal swabs

IPD SHARING:
Plan to Share IPD: Yes
all de-identified data would be available upon request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: within one month of request
Access Criteria: institutional approval